CLINICAL TRIAL: NCT02764528
Title: Effects of Promoting Handwashing With Soap to Improve Maternal Handwashing Behavior During the Neonatal Period
Brief Title: Intervention Study to Improve Maternal Handwashing
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Donor altered priorities for available funding and eliminated the project
Sponsor: State University of New York at Buffalo (Other)
Collaborators: Save the Children (Other); United States Agency for International Development (USAID) (U.S. Federal Agency); Unilever R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 748140-1; ESRC P176/2015 (Other: Amref)
Record Dates: First submitted 2016-01-13; First posted 2016-05-06 (Estimated); Last update posted 2022-09-23 (Actual); Status verified 2017-10

CONDITIONS: Infection; Neonatal
Keywords: Hygiene
MeSH Terms: conditions — Infections | interventions — Ambulatory Care Facilities; Home Care Services

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (No Intervention): Women will receive standard antenatal care but will not receive any additional handwashing promotion, soap, or handwashing device during their enrollment. At the end of data collection, handwashing with soap will be recommended to participants in the control arm and their families.
- Clinic (Experimental): Handwashing promotion from healthcare workers at antenatal care clinic.
  Interventions: Behavioral: Clinic
- Clinic + home (Experimental): Handwashing promotion from healthcare workers at antenatal care clinic and from community health volunteers at home visits.
  Interventions: Behavioral: Clinic + home
- Clinic + home + handwashing device (Experimental): Handwashing promotion from healthcare workers at antenatal care clinic and from community health volunteers at home visits with provision of one handwashing device.
  Interventions: Behavioral: Clinic + home + handwashing device

INTERVENTIONS:
Behavioral: Clinic — Pregnant women will receive handwashing promotion from a trained facility-based health care worker during her regular antenatal visit at a healthcare clinic. To the extent feasible, everyone accompanying the pregnant woman will be invited to take part in the behavior change communication session. The participant will be provided with several bars of soap to take home and she will be encouraged to maintain a designated place for washing hands (with soap and water) at the home. A poster indicating the key events for handwashing with soap will be posted at the clinic and smaller posters will be given to the participant to post in her home. A system will be established to send regular SMS messages to the participant promote handwashing with soap during the neonatal period.
  Arms: Clinic
Behavioral: Clinic + home — Women will receive all components of the clinic-based handwashing promotion in addition to handwashing promotion during 3-4 home visits before their expected delivery date and during the neonatal period from a community health volunteer. All household members present will be invited to join in the session, with emphasis on including all caregivers of the neonate.
  Arms: Clinic + home
Behavioral: Clinic + home + handwashing device — Women will receive all components of the clinic + home-based handwashing promotion intervention in addition to one handwashing device (i.e. tap and basin to use as a handwashing station) during the first home visit by the community health volunteer. The community health volunteer will work with the woman and her family to identify the location where the neonate will be most of the time in order to position the handwashing station as close to the neonate as possible.
  Arms: Clinic + home + handwashing device

SUMMARY:
The purpose of the handwashing intervention trial is to determine whether an interactive, storytelling approach to promoting handwashing with soap by health care workers can improve mothers' handwashing behavior during the first month of her child's life.

DETAILED DESCRIPTION:
Infectious diseases, such as umbilical cord infection, pneumonia, and sepsis, are responsible for about a quarter of neonatal deaths. Contaminated hands likely play a role in transmitting pathogens to a neonate, therefore handwashing with soap has the potential to interrupt transmission and improve neonatal health. The primary objective of this study is to develop and evaluate a scalable, cost-effective handwashing promotion program to improve handwashing behavior among mothers and caregivers of neonates. The investigators will first conduct a qualitative study to assess the feasibility and acceptability of a set of interventions. The investigators propose to evaluate the impact of the intervention components, designed as three progressively intense interventions, using a randomized controlled trial with elements of a stepped wedge design. The study will be conducted in Meru County, Kenya, enrolling a total of 800 pregnant women who seek non-emergency antenatal care at a government health facility during a 1 year period. Clinic based health care workers and community health volunteers will disseminate the intervention using an interactive storytelling approach. The focus of the interactions between the health care workers and volunteers and the participant will be on addressing barriers to handwashing through interactive question and answer sessions, rather than a didactic, educational session. The investigators will assess the impact of interventions on observed maternal and caregiver handwashing behavior and estimate the cost effectiveness for each intervention.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women
* Seeking routine (non-emergency) care at a participating antenatal care clinic during the study period
* Between 30 and 36 weeks pregnant (calculated based on last known menstrual period) when they seek antenatal care
* Live within 30 minutes or 1-2 km one-way travel from the clinic
* Plan to remain in the study area for at least one month post-partum
* Willing to allow the field worker to visit her home following the antenatal care visit on the day of enrollment to conduct baseline assessments at the household
* Sought antenatal care from a qualified medical provider for the first time at or after 28 weeks gestation

Exclusion Criteria:

* Excluded if another member of their household or compound/homestead enrolled in this study
* Excluded if enrolled in the formative research for this study

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-02-01 (Estimated); Primary Completion 2016-12-01 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Frequency of washing hands with soap at potential pathogen transmission events by mothers of neonate | 1 week post-natal
  Direct observation of handwashing behavior of mothers at times when pathogens may be transmitted from the mother to the neonate
Frequency of washing hands with soap at potential pathogen transmission events by mothers of neonate | 2 weeks post-natal
  Direct observation of handwashing behavior of mothers at times when pathogens may be transmitted from the mother to the neonate

SECONDARY OUTCOMES:
Frequency of washing hands with soap at potential pathogen transmission events by caregivers of neonate (other than mother) | 1 week post-natal
  Direct observation of handwashing behavior of caregivers (other than mother) at times when pathogens may be transmitted from the caregiver to the neonate
Number of participants with soap and water present at a handwashing station | 1 week post-natal
  Observed presence of soap and/or water at a handwashing station
Cost-effectiveness | 1 month post-partum
  Approximate cost of the intervention per participant
Frequency of washing hands with soap at potential pathogen transmission events by caregivers of neonate (other than mother) | 2 weeks post-natal
  Direct observation of handwashing behavior of caregivers (other than mother) at times when pathogens may be transmitted from the caregiver to the neonate
Number of participants with soap and water present at a handwashing station | 2 weeks post-natal
  Observed presence of soap and/or water at a handwashing station

CONTACTS AND LOCATIONS:
Overall Officials: Pavani K. Ram, M.D., Principal Investigator — State University of New York at Buffalo
Locations (1):
- Government funded antenatal care clinics, Igembe North and Igembe South Subcounties, Meru County, Kenya